CLINICAL TRIAL: NCT06775327
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled, Single-Dose, Dose Escalation, and Food-Effect Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Food Effect of INCB000631 When Administered Orally to Healthy Adult Participants
Brief Title: Study to Assess Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, & Food Effect of Oral INCB000631 to Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB000631-101
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Healthy Participants
Keywords: INCB000631

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort A (Experimental): INCB000631 or placebo will be administered at the protocol defined dose.
  Interventions: Drug: INCB000631; Drug: Placebo
- Cohort B (Experimental): INCB000631 or placebo will be administered at the protocol defined dose.
  Interventions: Drug: INCB000631; Drug: Placebo
- Cohort C (Experimental): INCB000631 or placebo will be administered at the protocol defined dose.
  Interventions: Drug: INCB000631; Drug: Placebo
- Cohort D (Experimental): INCB000631 or placebo will be administered at the protocol defined dose.
  Interventions: Drug: INCB000631; Drug: Placebo
- Cohort E (Experimental): INCB000631 or placebo will be administered at the protocol defined dose.
  Interventions: Drug: INCB000631; Drug: Placebo
- Optional Cohort F (Experimental): INCB000631 or placebo will be administered at the protocol defined dose.
  Interventions: Drug: INCB000631; Drug: Placebo
- Cohort G Treatment A (Experimental): INCB000631 will be administered at the protocol defined dose.
  Interventions: Drug: INCB000631
- Cohort G Treatment B (Experimental): INCB000631 will be administered at the protocol defined dose.
  Interventions: Drug: INCB000631

INTERVENTIONS:
Drug: INCB000631 — Oral; Tablet
Drug: Placebo — Oral; Tablet
  Arms: Cohort A; Cohort B; Cohort C; Cohort D; Cohort E; Optional Cohort F

SUMMARY:
This study will be conducted to assess the Safety, Tolerability, Pharmacokinetics (PK), Pharmacodynamics, and Food Effect of INCB000631 When Administered Orally to Healthy Adult Participants.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign a written ICF for the study.
* Aged 19 to 55 years, inclusive, at the time of signing the ICF.
* Body mass index between 18.0 and 32.0 kg/m2, inclusive, at screening. Note: Only up to 25% of the participants may be enrolled with a body mass index > 30 to ≤ 32.0 kg/m2.
* No clinically significant findings on screening evaluations (clinical, laboratory [except lipids], and ECG) as determined by the investigator. If the investigator has questions about clinically significant findings, the medical monitor should be consulted.
* Ability to swallow and retain oral tablets.
* Willingness to avoid pregnancy or fathering children based on the protocol defined criteria.

Exclusion Criteria:

* History of uncontrolled or unstable respiratory, renal, gastrointestinal, endocrine, pulmonary, hematopoietic, psychiatric, and/or neurological disease within 6 months of screening.
* History of an autoimmune disease (eg, myasthenia gravis).
* History of cardiovascular, cerebrovascular, cerebral, peripheral vascular, or thrombotic disease or uncontrolled hypertension.
* High blood pressure (systolic blood pressure > 140 mm Hg or diastolic blood pressure > 90 mm Hg at screening, confirmed by repeat testing).
* Confirmed resting pulse (up to 3 measurements) < 40 bpm or > 100 bpm at screening for vital signs.
* History or presence of an abnormal ECG before initial dose administration that, in the investigator's opinion, is clinically significant. Participants with a QTcF interval > 450 milliseconds (males) or > 470 milliseconds (females), QRS interval > 120 milliseconds, or PR interval > 220 milliseconds will be excluded.

In the event a value is exclusionary, a single ECG will be repeated twice, and an average of the 3 readings will be used to determine if a participant should be excluded.

* Presence or history of a malabsorption syndrome possibly affecting drug absorption (eg, Crohn disease or chronic pancreatitis).
* History of malignancy within 5 years of screening, with the exception of cured basal cell or squamous cell carcinoma of the skin, ductal carcinoma in situ, or Gleason 6 prostate cancer.
* History of other malignancy within 2 years of screening (with the exception of cured basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy) or cancers from which the participant has been disease-free for < 1 year after treatment with curative intent.
* Current or recent (within 3 months of screening) clinically significant gastrointestinal disease or surgery (including cholecystectomy; excluding appendectomy and hernia repair) that could affect the absorption of study drug.
* Hemoglobin, WBC count, platelet count, or absolute neutrophil count less than the laboratory lower limit of normal at screening or at check-in, confirmed by repeat testing, that is considered clinically significant in the opinion of the investigator to be exclusionary.
* Hepatic transaminases (ALT and AST), ALP, or total bilirubin > 1.25 × the laboratory-defined ULN at screening or at check-in, confirmed by repeat testing (except participants with Gilbert disease, for whom total bilirubin must be ≤ 2.0 × ULN).
* Any major surgery within 4 weeks of screening.
* Donation of blood to a blood bank or participation in a clinical study (except a screening visit) within 4 weeks of screening (within 2 weeks for donation of plasma only).
* Blood transfusion within 4 months of check-in (Day -1).
* Chronic, known, or current active infectious disease requiring systemic antibiotic, antifungal, or antiviral treatment (includes latent tuberculosis).
* Positive test for HBV, HCV, or HIV. Participants whose results are compatible with prior immunization for or immunity due to infection with HBV may be included at the discretion of the investigator.
* Received a live vaccine (including attenuated) within 3 months of the planned start of the study drug or anticipation of need for such a vaccine during the study. This includes seasonal influenza vaccines.

Note: Examples of live vaccines include but are not limited to the following: measles, mumps, rubella, chickenpox/zoster, yellow fever, rabies, Bacillus Calmette-Guérin, and typhoid.

* History of significant alcohol use within 3 months of screening, defined as regular alcohol consumption > 21 units per week for males and > 14 units for females (1 unit = one-half pint of beer or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine).
* Positive urine or breath test for ethanol or positive urine or serum screen for drugs of abuse that are not otherwise explained by permitted concomitant medications or diet.
* Ingestion of caffeine- or xanthine-containing products (eg, coffee, tea, cola drinks, energy drinks, and chocolate) within 48 hours before check-in.
* Consumption of alcoholic beverages, Seville oranges, grapefruit or grapefruit juice, pomelos, exotic citrus fruits, grapefruit hybrids, or fruit juices within 48 hours before check-in.
* History of tobacco or nicotine-containing product use within 1 month of screening.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before the first dose of study drug with another investigational medication or current enrollment in another investigational drug study.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before the first dose of study drug with an inducer or inhibitor of CYP3A4, P-gp, or BCRP (refer to the Certara Drug Interaction Database for prohibited drugs).
* Current use of prohibited medication as described in the protocol.
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity) deemed clinically relevant by the investigator.
* Known hypersensitivity or severe reaction to INCB000631 or any excipients of INCB000631 or any SPPL2a inhibitors (refer to the IB).
* Inability to undergo venipuncture or tolerate venous access (participant has inadequate veins for repeat venipuncture or venous access as determined by the investigator or designee).
* Inability or unlikeliness of the participant to comply with the dose schedule and study evaluations, in the opinion of the investigator or designee.
* Use of prescription drugs (including hormonal contraceptives) within 14 days of study drug administration or nonprescription medications/products (including minerals and phytotherapeutics/herbals [including St John's wort]/plant-derived preparations) within 7 days of study drug administration. However, occasional and standard-dose acetaminophen and standard-dose vitamins are permitted. Mega-dose vitamins or supplements are not permissible.
* Pregnant or breastfeeding.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* eGFR < 90 mL/min/1.73 m2 based on the site's standard formula at screening. Note: Assessment of eGFR may be repeated once if outside of the reference range.
* Excessive exercise beyond the activities of daily living (eg, triathlon) within 7 days before check-in (Day -1).
* History of severe lactose intolerance or food allergies/intolerance to the composition of the standard high-fat breakfast to be served (Cohort G only).

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2025-02-13 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to Day 41
  Defined as any adverse event, either reported for the first time or the worsening of a pre-existing event, occurring after dose of study treatment.
PK for plasma INCB000631: Cmax | Up to Day 14
  Maximum Observed Plasma Concentration of INCB000631.
PK for plasma INCB000631: tmax | Up to Day 14
  Time to maximum plasma concentration of INCB000631.
PK for plasma INCB000631: AUC(0-t) | Up to Day 14
  Area under the single-dose plasma concentration-time curve up to the last measurable plasma concentration of INCB000631.
PK for plasma INCB000631: AUC 0-∞ | Up to Day 14
  Area under the single-dose plasma concentration-time curve from 0 to Infinity of INCB000631.

SECONDARY OUTCOMES:
PK for plasma INCB000631: t1/2 | Up to Day 14
  Apparent terminal phase disposition half-life of INCB000631.
PK for plasma INCB000631: CL/F | Up to Day 14
  Dose clearance of INCB000631.
PK for plasma INCB000631: Vz/F | Up to Day 14
  Apparent oral dose volume of distribution of INCB000631.
PK for plasma INCB000631: λz | Up to Day 14
  Apparent terminal-phase disposition rate constant of INCB000631.
PK for urine INCB000631: Ae96h | Up to Day 14
  Amount of INCB000631 excreted in the urine over 96 hours.
PK for urine INCB000631: fe | Up to Day 14
  Percent of INCB000631 excreted in the urine.
PK for urine INCB000631: CLR | Up to Day 14
  Renal clearance of INCB000631.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (1):
- Celerion, Inc, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study to Assess Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, & Food Effect of Oral INCB000631 to Healthy Adult Participants — https://www.incyteclinicaltrials.com/study/?id=INCB000631-101&SearchTerm=INCB000631-101&Latitude=&Longitude=&LocationName=&conditions=&Status=&phases=&AgeRanges=&gender=&StudyTypes=&AttachmentTypes=&MileRadius=100&PageIndex=0&PageSize=10&SortField=&SortOrder=&hasResults=